CLINICAL TRIAL: NCT04654858
Title: Restoration of Permanent Molars Affected With Molar-incisor-hypomineralization (MIH) Among a Group of Egyptian Children Using Composite Restorations or Preformed Metal Crowns: Two-arm Randomized Controlled Trial (Part II)
Brief Title: Restoration of Permanent Molars Affected With (MIH) Using Composite Restorations or Preformed Metal Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amal Ahmed Mohamed El Kot (Other)
Responsible Party: Sponsor-Investigator, Amal Ahmed Mohamed El Kot, doctor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: treatment of teeth with MIH
Record Dates: First submitted 2020-11-03; First posted 2020-12-04 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Molar Incisor Hypomineralization
Keywords: MIH
MeSH Terms: conditions — Molar Hypomineralization | interventions — Composite Resins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding to the child participants and legal guardian of each participating child, operator, outcome assessor and statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct composite restorations (Active Comparator): bulk-fill composite (Filtek BulkFlow, 3M Espe) will be used after infiltration or block anaesthesia for affected molar, following by carious tissue removal. Marginal bevelling of enamel will be performed. A universal adhesive (Scotchbond Universal, 3M Espe) will be placed after selective enamel etching A bulk-fill composite will be used and covered using a nanohybrid composite, (Filtek XT, 3M Espe).
  Interventions: Procedure: Direct composite restorations
- Performed metal crowns (Active Comparator): PMCs (3M Espe, Seefeld, Germany) will be placed after infiltration or block anaesthesia for affected molar, followed by removal of carious dentin and enamel, Tooth preparation for fitting the crown, The correct size of crown will be chosen, and then Cemented with glass ionomer luting cement (KetacCem, 3M Espe).
  Interventions: Procedure: Direct composite restorations

INTERVENTIONS:
Procedure: Direct composite restorations — bulk-fill composite (Filtek BulkFlow, 3M Espe) will be used aftar infiltration or block anaesthesia for affected molar,following by carious tissue removal. Marginal bevelling of enamel will be performed. A universal adhesive (Scotchbond Universal, 3M Espe) will be placed after selective enamel etching A bulk-fill composite will be used and covered using a nanohybrid composite, (Filtek XT, 3M Espe).
  Other Names: composite resin

SUMMARY:
The aim of this study is to compare the clinical outcome of using direct esthetic composite restorations in managing MIH cases and the use of preformed metal crowns.

DETAILED DESCRIPTION:
Molar incisor hypomineralization can represent a serious and challenging clinical management problem. Children with MIH require higher levels of treatment needs and demonstrate considerable management problems.

For most severely affected MIH molars, direct esthetic restorative materials or preformed metal crowns will be the treatments to choose between. A number of aspects which could support decision-making, however, are not clearly demarcated. First and foremost, it is not clear if both treatments are similarly acceptable for patients and providers.

ELIGIBILITY:
Inclusion Criteria:

1. Children with MIH in one fully erupted molar or more.
2. Age ranging from 7-12 years.
3. cooperative children
4. Good general health.

Exclusion Criteria:

1. patients participating in other experiments.
2. Patients with parents planning to move away within the following year.
3. Patients with only mildly affected MIH molars that do not require extensive restorative treatment.
4. MIH-affected molars that have a very poor prognosis and require extraction.
5. First permanent molars that are affected with other developmental defects, such as hypoplasia, dental fluorosis or amelogenesis imperfecta.

   -

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-07-04 (Actual); Primary Completion 2023-09-03 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
Hypersensitivity | 12 month
  Questioning the patient and/or the parent (Clemenus et al,2017) Binary (yes, no)

SECONDARY OUTCOMES:
Acceptability of the treatment | 12 month
  Questioning the children or parents about accepting the treatment Binary (Yes or No)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] • • Alanzi A, Faridoun A, Kavvadia K, Ghanim A. 2018. Dentists' perception, knowledge, and clinical management of molar-incisor-hypomineralisation in kuwait: A cross-sectional study. BMC oral health. 18(1):34. • Bakkal M, Abbasoglu Z, Kargul B. 2017. The effect of casein phosphopeptide-amorphous calcium phosphate on molar-incisor hypomineralisation: A pilot study. Oral health & preventive dentistry. 15(2):163-167. • Baroni C, Marchionni S. 2011. Mih supplementation strategies: Prospective clinical and laboratory trial. Journal of dental research. 90(3):371-376. • Bekes K, Heinzelmann K, Lettner S, Schaller HG. 2016. Efficacy of desensitizing products containing 8% arginine and calcium carbonate for hypersensitivity relief in mih-affected molars: An 8-week clinical study. Clinical oral investigations. • Bekes K, Steffen R. 2016. Das würzburger mih - konzept: Teil 1. Der mih - treatment need index (mih - tni). Ein neuer index zur befunderhebung und therapieplanung bei patienten mit molaren - inzisiven hypomineralisation Oralprophylaxe & Kinderzahnheilkunde. 38(4):165-170. • Briggs A, Sculpher M. 1997. Commentary: Markov models of medical prognosis. BMJ. 314 (7077):345-345.Briggs AH, O'Brien BJ, Blackhouse G. 2002. Thinking outside the box: Recent advances in the analysis and presentation of uncertainty in cost-effectiveness studies. Annual Review of Public Health. 23(1):377-401. • Byford, S., Knapp, M., Greenshields, J., Byford, S., Knapp, M., Greenshields, J., et al (2003) Cost-effectiveness of brief cognitive behaviour therapy Cost-effectiveness of brief cognitive behaviour therapy versus treatment as usual in recurrent deliberate self- versus treatment as usual in recurrent deliberate selfharm: a rational decision making approach. harm: a rational decision making approach. Psychological Psychological MedicineMedicine, 33, 977 • Cuzick J. 2005. Rank regression. Encyclopedia of biostatistics vol 6. Wiley and Sons. de Souza JF, Fragelli CB, Jeremias F, Paschoal MAB, Santos-Pinto L, de Cassia Loiola Cordeiro R. 2017. • Eighteen-month clinical performance of composite resin restorations with two different adhesive systems for molars affected by molar incisor hypomineralization. Clinical oral investigations. 21(5):1725-1733. • Dworkin SL. 2012. Sample size policy for qualitative studies using in-depth interviews. Archives of sexual behavior. 41(6):1319-1320. • Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA. 2016. Consort 2010 statement: Extension to randomised pilot and feasibility trials. Bmj. 355:i5239